CLINICAL TRIAL: NCT00545272
Title: A Randomized, Multi-center, Parallel Group, Double Blind, Placebo and Formoterol Controlled 14 Day Dose Ranging Trial of 4 Doses of Indacaterol Delivered Via TWISTHALER® Device in Adult and Adolescent Patients With Persistent Asthma
Brief Title: A Dose Ranging Trial of 4 Doses of Indacaterol Delivered Via TWISTHALER® Device in Adult and Adolescent Patients With Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQMF149A2201; 2007-003191-19 (EudraCT Number)
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2012-11

CONDITIONS: Asthma
Keywords: QMF; indacaterol; Twisthaler®
MeSH Terms: conditions — Asthma | interventions — indacaterol; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- indacaterol 62.5 μg (Experimental): Indacaterol 62.5 μg delivered by the TWISTHALER® device once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days. All participants were supplied with salbutamol/albuterol to use throughout the study as rescue medication.
  Interventions: Drug: indacaterol; Drug: placebo to formoterol; Drug: short acting β2-agonist
- indacaterol 125 μg (Experimental): Indacaterol 125 μg delivered by the TWISTHALER® device once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days. All participants were supplied with salbutamol/albuterol to use throughout the study as rescue medication.
  Interventions: Drug: indacaterol; Drug: placebo to formoterol; Drug: short acting β2-agonist
- indacaterol 250 μg (Experimental): Indacaterol 250 μg delivered by the TWISTHALER® device once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days. All participants were supplied with salbutamol/albuterol to use throughout the study as rescue medication.
  Interventions: Drug: indacaterol; Drug: placebo to formoterol; Drug: short acting β2-agonist
- indacaterol 500 μg (Experimental): Indacaterol 500 μg delivered by the TWISTHALER® device once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days. All participants were supplied with salbutamol/albuterol to use throughout the study as rescue medication.
  Interventions: Drug: indacaterol; Drug: placebo to formoterol; Drug: short acting β2-agonist
- formoterol (Active Comparator): Formoterol 12 μg delivered by the AEROLIZER® device twice a day and placebo to indacaterol (placebo TWISTHALER® device) once a day for 14 days. All participants were supplied with salbutamol/albuterol to use throughout the study as rescue medication.
  Interventions: Drug: formoterol; Drug: placebo to indacaterol; Drug: short acting β2-agonist
- placebo (Placebo Comparator): Placebo to indacaterol (placebo TWISTHALER® device) once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days. All participants were supplied with salbutamol/albuterol to use throughout the study as rescue medication.
  Interventions: Drug: placebo to indacaterol; Drug: placebo to formoterol; Drug: short acting β2-agonist

INTERVENTIONS:
Drug: indacaterol — Indacaterol delivered by multiple dose dry powder inhaler (TWISTHALER® device).
  Arms: indacaterol 125 μg; indacaterol 250 μg; indacaterol 500 μg; indacaterol 62.5 μg
Drug: formoterol — Formoterol delivered by oral inhalation via AEROLIZER® inhalation device.
  Arms: formoterol
Drug: placebo to indacaterol — Placebo TWISTHALER® device
  Arms: formoterol; placebo
Drug: placebo to formoterol — Placebo AEROLIZER® device
  Arms: indacaterol 125 μg; indacaterol 250 μg; indacaterol 500 μg; indacaterol 62.5 μg; placebo
Drug: short acting β2-agonist — 100 μg/ 90 μg salbutamol/albuterol Metered Dose Inhaler (MDI) or equivalent dose of Dry Powder Inhaler (DPI).

SUMMARY:
This study will evaluate the dose response relationship among four doses of indacaterol as well as placebo delivered via the TWISTHALER® device.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adult and adolescent patients aged 12-75 years inclusive (or ≥18-75 years depending upon regulatory and/or Institutional Review Board (IRB)/Independent Ethics Committee (IEC)/Research Ethics Board (REB) approval), who have signed an Informed Consent Form prior to initiation of any study-related procedure, including any adjustments to asthma medication prior to Visit 1. Patients below the legal age of consent are required to have the Informed Consent Form signed by the patient's parent / guardian.
2. Patients with asthma, diagnosed according to Global Initiative for Asthma (GINA) guidelines (National Institute of Health, National Heart, Lung and Blood Institute, 2006) and who additionally meet the following criteria:

   1. Patients receiving daily treatment with inhaled corticosteroid up to the maximum dose per day indicated in the package leaflet, in a stable regimen for the month prior to Visit 1.
   2. Patients with a Forced Expiratory Volume in one second (FEV1) at Visit 1 of ≥50% of the predicted normal value for the patient. This criterion for FEV1 will have to be demonstrated after a washout period of at least 6 hours during which no short acting β2-agonist has been inhaled, and a minimum of 48 hours for a long acting β2-agonist.
   3. Patients who demonstrate an increase of ≥12% and ≥200 mL in FEV1 over their pre-bronchodilator value within 30 minutes after inhaling a total of 200 µg/180 µg of salbutamol/albuterol Metered Dose Inhaler (MDI) (or equivalent dose of Dry Powder Inhaler [DPI]) (the reversibility test). Reversibility will have to be demonstrated after an appropriate washout period of at least 6 hrs prior to the evaluation for a short-acting β2-agonist. The administration of salbutamol/albuterol for the reversibility test is to be within 30 minutes after pre bronchodilator spirometry. Reversibility has to be demonstrated at Visit 1 or between Visits 1 and 2, in order for patients to be included in the trial.

Exclusion Criteria:

* Pregnant women, nursing mothers, or females of childbearing potential, regardless of whether or not sexually active, if they are not using a reliable form of contraception.
* Patients with Chronic Obstructive Pulmonary Disease (COPD), or current smokers, or patients who have used tobacco products within the 6 month period prior to Visit 1, or who have a smoking history of greater than 10 pack years.
* Patients:

  1. who's asthma is likely to deteriorate during the study (including seasonal allergy),
  2. hospitalized for an acute asthma attack/asthma exacerbation within 6 months prior to Visit 1,
  3. who have had an emergency room visit for an asthma attack/asthma exacerbation within 6 weeks prior to Visit 1
  4. who have had a respiratory tract infection or emergency room treatment for an asthma attack/asthma exacerbation within 4 weeks prior to Visit 1
  5. Patients who require the use of ≥8 inhalations per day of short acting B2-agonist (100 µg/ 90 µg salbutamol/albuterol MDI or equivalent dose of DPI) on any 2 consecutive days from Screening to Randomization.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2007-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma, Study Chair — Novartis Pharmaceuticals
Locations (60):
- Belgium (4):
  - Novartis Investigator Site, Aalst
  - Novartis Investigator Site, Halen
  - Novartis Investigator Site, Oostham
  - Novartis Investigator site, Veurne
- Czechia (6):
  - Novartis Investigator Site, Boskovice
  - Novartis Investigator Site, Brno
  - Novartis Investigator site, Břeclav
  - Novartis Investigator Site, Liberec
  - Novartis Investigator Site, Most
  - Novartis Investigator Site, Tábor
- Germany (7):
  - Novartis Investigator Site, Aalen
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Braunschweig
  - Novartis Investigator Site, Deggendorf
  - Novartis Investigator Site, Fürstenwalde
  - Novartis Investigator Site, Leipzig
  - novartis Investigator site, München
- Hungary (8):
  - Novartis investigator site, Balassagyarmat
  - Novartis Investigator Site, Érd
  - Novartis Investigator site, Füzesabony
  - Novartis Investigator Site, Gyonggyos
  - Novartis Investigator Site, Mosdoz
  - Novartis Investigator Site, Pest
  - Novartis Investigator Site, Siófok
  - Novartis Investigator Site, Százhalombatta
- Israel (10):
  - Novartis Investigator Site, Afula
  - Novartis Investigator Site, Ashkelon
  - Novartis Investigator Site, Beersheba
  - Novartis investigator site, Haifa
  - Novartis investigator site, Jerusalem
  - Novartis Investigator Site, Petah Tikva
  - Novartis Investigator Site, Rehovot
  - Novartis Investigator Site, Tel Aviv
  - Novartis Investigator Site, Tel-Hashorner
  - Novartis Investigator Site, Zrifin
- Poland (5):
  - Novartis Investigator Site, Bialystok
  - Novartis investigator site, Bydgoszcz
  - Novartis Investigator Site, Lodz
  - Novartis Investigator site, Lubin
  - Novartis Investigator Site, Tarnów
- Russia (4):
  - Novartis Investigator Site, Moscow
  - Novartis Investigator Site, Saint Petersburg
  - Novartis Investigator Site, Smolensk
  - Novartis investigator site, Tomsk
- South Africa (8):
  - Novartis Investigator Site, Bloernfontain
  - Novartis Investigator Site, Cape Town
  - Novartis Investigator Site, Johannesburg
  - Novartis Investigator Site, Krugersdorp
  - Novartis Investigator Site, Les Marais
  - Novartis Investigator Site, Pretoria
  - Novartis Investigator Site, Roodepoort
  - Novartis Investigator Site, Themba
- Spain (3):
  - Novartis Investigator Site, Madrid
  - Novartis Investigator Site, Pozuelo de Alacron
  - Novartis Investigator Site, Valencia
- United Kingdom (5):
  - Novartis Investigator Site, Downpatrick
  - Novartis Investigator Site, Glasgow
  - Novartis Investigator Site, London
  - Novartis Investigator Site, Southampton
  - Novartis Investigator Site, Watford

RESULTS

PARTICIPANT FLOW:
Groups:
- Indacaterol 62.5 μg: Indacaterol 62.5 μg delivered by the TWISTHALER® device once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days.
- Indacaterol 125 μg: Indacaterol 125 μg delivered by the TWISTHALER® device once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days.
- Indacaterol 250 μg: Indacaterol 250 μg delivered by the TWISTHALER® device once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days.
- Indacaterol 500 μg: Indacaterol 500 μg delivered by the TWISTHALER® device once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days.
- Formoterol: Formoterol 12 μg delivered by the AEROLIZER® device twice a day and placebo to indacaterol (placebo TWISTHALER® device) once a day for 14 days.
- Placebo: Placebo to indacaterol (placebo TWISTHALER® device) once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days.
Period: Overall Study
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Started | 61 | 68 | 65 | 72 | 64 | 62
Completed | 61 | 67 | 64 | 71 | 62 | 59
Not Completed | 0 | 1 | 1 | 1 | 2 | 3
Not completed — Protocol deviation | 0 | 1 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Abnormal laboratory value(s) | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Abnormal test procedure result(s) | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo | Total
Number analyzed (Participants) | 61 | 68 | 65 | 72 | 64 | 62 | 392
Age Continuous [Mean (Standard Deviation); unit: years] | 41.3 (16.27) | 38.4 (17.25) | 36.6 (15.76) | 40.1 (15.47) | 44.0 (17.98) | 39.8 (15.82) | 40.0 (16.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 37 | 36 | 39 | 27 | 37 | 204
  Male | 33 | 31 | 29 | 33 | 37 | 25 | 188

OUTCOME MEASURES:

1. Primary Outcome: The Mean Change From Baseline to 24 Hour Post-dose (Trough) Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Change from baseline to 24 hour post dose trough FEV1 after 14 days of treatment was analyzed using Analysis of Covariance (ANCOVA) adjusting for treatment and region with baseline FEV1 as a covariate.
Time Frame: Baseline (prior to first dose) and Day 15 (24 hours after last dose)
Population: The intent-to-treat population (ITT) population consisted of all randomized patients who had a baseline and at least one post-dose FEV1 measurement. The analysis only includes patients with non-missing data.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Number analyzed (Participants) | 60 | 67 | 63 | 68 | 62 | 58
liters | 0.039 (0.0408) | 0.054 (0.0383) | 0.124 (0.0401) | 0.166 (0.0381) | 0.075 (0.0405) | -0.018 (0.0415)

2. Secondary Outcome: Standardized Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC) Between Baseline (Predose) and 4 Hours Post-dose
Description: FEV1 was measured on Day 14 pre-dose and up to 4 hours post-dose. The Area Under the Curve (AUC) for FEV1 was analyzed using Analysis of Covariance adjusting for treatment and region with baseline FEV1 as a covariate.
Time Frame: Day 14, pre-dose, 5, 20 and 30 minutes, 1, 2, 3, and 4 hours post-dose.
Population: The intent-to-treat population (ITT) population consisted of all randomized patients who had a baseline and at least one post-dose FEV1 measurement. Observed data only.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Number analyzed (Participants) | 61 | 66 | 64 | 69 | 62 | 59
liters | 2.670 (0.0419) | 2.698 (0.0400) | 2.772 (0.0411) | 2.786 (0.0393) | 2.821 (0.0418) | 2.565 (0.0426)

3. Secondary Outcome: The Mean Change From Baseline to 24 Hour Post-dose (Trough) Forced Expiratory Volume in 1 Second (FEV1) on Day 1
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Change from baseline to 24 hour post dose trough FEV1 after 1 day of treatment was analyzed using Analysis of Covariance (ANCOVA) adjusting for treatment and region with baseline FEV1 as a covariate.
Time Frame: Day 1 Baseline (prior to first dose) and 24 hours post-dose.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Number analyzed (Participants) | 61 | 68 | 64 | 69 | 63 | 62
liters | 0.054 (0.0347) | 0.081 (0.0326) | 0.143 (0.0339) | 0.141 (0.0326) | 0.155 (0.0341) | 0.010 (0.0344)

4. Secondary Outcome: Standardized Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC) Between Baseline (Predose) and 4 Hours Post-dose on Day 1
Description: FEV1 was measured on Day 1 pre-dose and up to 4 hours post-dose. The Area Under the Curve (AUC) for FEV1 was analyzed using Analysis of Covariance adjusting for treatment and region with baseline FEV1 as a covariate.
Time Frame: Day 1, pre-dose, 5, 20 and 30 minutes, 1, 2, 3, and 4 hours post-dose.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Number analyzed (Participants) | 61 | 68 | 65 | 71 | 64 | 62
liters | 2.668 (0.0281) | 2.687 (0.0264) | 2.726 (0.0272) | 2.753 (0.0259) | 2.832 (0.0274) | 2.547 (0.0279)

5. Secondary Outcome: Time to Peak Forced Expiratory Volume in 1 Second (FEV1) on Day 1 and Day 14
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Time to peak FEV1 is calculated in minutes from the time of inhalation of study drug to the time of the peak FEV1, which is taken as the maximum FEV1 recorded post-dose.
Time Frame: Day 1 and Day 14 measured pre-dose and up to 4 hours post-dose
Population: The intent-to-treat population (ITT) population consisted of all randomized patients who had a baseline and at least one post-dose FEV1 measurement. The analysis only includes patients with non-missing data, indicated by "N".
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Number analyzed (Participants) | 61 | 68 | 65 | 72 | 64 | 62
minutes
  Day 1 [N=61, 68, 65, 71, 64, 62] | 91.0 (83.02) | 109.6 (81.09) | 119.0 (81.64) | 116.2 (75.50) | 105.6 (70.64) | 90.5 (82.46)
  Day 14 [N=61, 66, 64, 70, 62, 59] | 103.8 (86.67) | 118.7 (88.42) | 96.7 (70.65) | 114.0 (76.41) | 114.6 (71.64) | 80.4 (76.92)

6. Secondary Outcome: Change From Baseline in Morning and Evening Peak Expiratory Flow
Description: The Peak Expiratory Flow (PEF) rate is the maximal rate that a person can exhale during a short maximal expiratory effort after fully inhaling. Participants measured their PEF using a peak flow meter and recorded measurements in a diary every morning and evening during the study, prior to taking study medication. Change from baseline is the difference between the mean baseline PEF recorded during the screening period until the first day of treatment, and the overall mean PEF from Days 1 to 14.
Time Frame: Baseline (recorded during the screening period) and Days 1-14 (treatment period)
Population: Intent to treat population. The analysis only includes patients with non-missing data, indicated by "N".
Measure: Mean (Standard Deviation); unit: liters/minute
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Number analyzed (Participants) | 61 | 68 | 65 | 72 | 64 | 62
liters/minute
  Morning [N=56, 61, 53, 63, 57, 48] | 18.7 (29.28) | 17.2 (34.07) | 25.7 (38.37) | 25.8 (47.36) | 25.2 (38.28) | -4.3 (43.00)
  Evening [N=56, 58, 54, 59, 55, 47] | 5.9 (36.92) | 4.2 (37.82) | 18.4 (36.70) | 25.8 (38.07) | 26.2 (35.01) | -11.4 (50.73)

7. Secondary Outcome: Number of Participants Using Rescue Medication
Description: Participants recorded the use of rescue medications (salbutamol/albuterol) for treatment of asthma symptoms twice a day in a diary during the 14 days of the treatment period.
Time Frame: Over 14 days
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Number analyzed (Participants) | 61 | 68 | 65 | 72 | 64 | 62
participants
  Night | 36 | 40 | 36 | 34 | 31 | 40
  Day | 33 | 43 | 28 | 35 | 30 | 39

ADVERSE EVENTS:
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/68 | 0/65 | 0/72 | 0/64 | 1/62
Other Adverse Events (participants affected / at risk) | 2/61 | 2/68 | 4/65 | 8/72 | 0/64 | 1/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 62.5 μg (N=61) | Indacaterol 125 μg (N=68) | Indacaterol 250 μg (N=65) | Indacaterol 500 μg (N=72) | Formoterol (N=64) | Placebo (N=62)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 62.5 μg (N=61) | Indacaterol 125 μg (N=68) | Indacaterol 250 μg (N=65) | Indacaterol 500 μg (N=72) | Formoterol (N=64) | Placebo (N=62)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4 | 8 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.